CLINICAL TRIAL: NCT06808087
Title: Comparison of the Efficacy of Transversus Abdominis Plane Block and Erector Spinae Plane Block in the Management of Acute Appendicitis Pain in the Emergency Department
Brief Title: Management of Acute Appendicitis Pain in the Emergency Department
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: AEŞH-EK1-2024-0037
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Acute Appendicitis
Keywords: Transversus Abdominis Plane Block; Erector Spinae Plane Block; Acute Appendicitis; Pain Management; Emergency Department
MeSH Terms: conditions — Appendicitis; Agnosia; Emergencies | interventions — Tramadol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T-50: Patients in the T-50 group will receive a 100 cc isotonic 0.9% NaCl (normal saline) solution containing 50 mg tramadol as an intravenous infusion over 15 minutes at baseline.
  Interventions: Drug: Tramadol
- TAP-50: Patients in the TAP-50 group will receive the same intravenous tramadol infusion as the T-50 group at baseline, followed by a TAP block.
  Interventions: Procedure: Transversus abdominis plane blockage; Drug: Tramadol
- ESPB-50: Patients in the ESPB-50 group will receive the same intravenous tramadol infusion as the T-50 group at baseline, followed by an ESP block.
  Interventions: Procedure: Erector spinae plane blockage; Drug: Tramadol

INTERVENTIONS:
Procedure: Transversus abdominis plane blockage — 1. Patient monitoring
  2. Preparation of the skin with 10% povidone-iodine and ensuring appropriate draping
  3. Placement of a high-frequency linear transducer transversely between the right iliac crest and subcostal margin along the midaxillary line. Structures visualized on ultrasound from superficial to deep include: skin, subcutaneous fat, external oblique muscle, internal oblique muscle, transversus abdominis muscle, and peritoneum. The TAP block will be performed in the transversus abdominis plane (TAP) between the internal oblique and transversus abdominis muscles.
  4. A 23-gauge, 60 mm blunt-tipped needle will be directed toward the TAP, and negative aspiration will be confirmed upon entry into the fascial layer.
  5. An injection of 20 mL of 0.25% bupivacaine, prepared by diluting 10 mL of 0.5% bupivacaine with 10 mL of normal saline, will be performed.
  6. Visualization of the oval spread of bupivacaine in the TAP.
  Groups: TAP-50
Procedure: Erector spinae plane blockage — 1. Patient monitoring
  2. Positioning the patient in the prone position
  3. Preparation of the skin with 10% povidone-iodine and ensuring appropriate draping
  4. Counting the transverse processes from the sacrum to find the L1 level
  5. Placing a low-frequency curvilinear transducer (depth set to 3-5 cm) parasagittally, and identifying the tip of the right transverse process at this level
  6. Visualizing the erector spinae muscle overlying the transverse process
  7. Inserting a 22G, 80 mm needle between the transverse process and the fascia of the erector spinae muscle
  8. Injecting 1 to 3 mL of saline to confirm the separation of the erector spinae muscle fascia from the transverse process after negative aspiration
  9. Injecting 20 mL of 0.25% bupivacaine, prepared by diluting 10 mL of 0.5% bupivacaine with 10 mL of normal saline, after another negative aspiration
  10. Visualizing the oval spread of bupivacaine over the erector spinae muscle.
  Groups: ESPB-50
Drug: Tramadol — 50 mg of tramadol will be administered via IV infusion over 15 minutes in 100 cc of isotonic 0.9% NaCl (normal saline).

SUMMARY:
This study aims to compare the effectiveness of TAP block, ESP block, and tramadol in preoperative pain management for patients diagnosed with acute appendicitis and undergoing emergency surgery in the emergency department. The study will evaluate the potential of TAP block and ESP block administered to patients diagnosed with acute appendicitis in the emergency department to reduce pain intensity before surgical intervention. With this study, we aim to contribute to practical applications to ensure optimal pain control for acute appendicitis patients under emergency department conditions.

DETAILED DESCRIPTION:
Our study will include patients who present to the emergency department with abdominal pain, receive a diagnosis of acute appendicitis through history, physical examination, and imaging modalities, and are determined to undergo definitive surgery following general surgical consultation. Patients will be randomly assigned to three groups. Randomization will be achieved by allocating the first 5 patients to the T-50 group, the second 5 patients to the TAP-50 group, and the third 5 patients to the ESPB-50 group. Patients' pain levels will be assessed using the Numeric Rating Scale (NRS) at baseline. Subsequently, patients in the T-50 group will receive a 100 cc isotonic 0.9% NaCl (normal saline) solution containing 50 mg tramadol as an intravenous infusion over 15 minutes at baseline. Patients in the TAP-50 group will receive the same intravenous tramadol infusion as the T-50 group at baseline, followed by a transversus abdominis plane (TAP) block. The steps for performing the TAP block are as follows:

1. Patient monitoring
2. Preparation of the skin with 10% povidone-iodine and ensuring appropriate draping
3. Placement of a high-frequency linear transducer transversely between the right iliac crest and subcostal margin along the midaxillary line. Structures visualized on ultrasound from superficial to deep include: skin, subcutaneous fat, external oblique muscle, internal oblique muscle, transversus abdominis muscle, and peritoneum. The TAP block will be performed in the transversus abdominis plane (TAP) between the internal oblique and transversus abdominis muscles.
4. A 23-gauge, 60 mm blunt-tipped needle will be directed toward the TAP, and negative aspiration will be confirmed upon entry into the fascial layer.
5. An injection of 20 mL of 0.25% bupivacaine, prepared by diluting 10 mL of 0.5% bupivacaine with 10 mL of normal saline, will be performed.
6. Visualization of the oval spread of bupivacaine in the TAP.

Patients in the ESPB-50 group will receive a 100 cc isotonic 0.9% NaCl (normal saline) solution containing 50 mg tramadol as an intravenous infusion over 15 minutes at baseline, followed by an ESP block. The steps for performing the ESP block are as follows:

1. Patient monitoring
2. Positioning the patient in the prone position
3. Preparation of the skin with 10% povidone-iodine and ensuring appropriate draping
4. Counting the transverse processes from the sacrum to find the L1 level
5. Placing a low-frequency curvilinear transducer (depth set to 3-5 cm) parasagittally, and identifying the tip of the right transverse process at this level
6. Visualizing the erector spinae muscle overlying the transverse process
7. Inserting a 22G, 80 mm needle between the transverse process and the fascia of the erector spinae muscle
8. Injecting 1 to 3 mL of saline to confirm the separation of the erector spinae muscle fascia from the transverse process after negative aspiration
9. Injecting 20 mL of 0.25% bupivacaine, prepared by diluting 10 mL of 0.5% bupivacaine with 10 mL of normal saline, after another negative aspiration
10. Visualizing the oval spread of bupivacaine over the erector spinae muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients who provide written consent

Exclusion Criteria:

* Patients with abdominal wall anatomical abnormalities
* Patients with known local anesthetic allergies
* Patients with a BMI >30
* Patients weighing less than 45 kg
* Patients with coagulopathy
* Patients with opioid, alcohol, or substance dependence
* Patients with skin infections at the site of local anesthetic administration
* Pregnant or breastfeeding patients
* Hemodynamically unstable patients
* Patients with liver or kidney failure
* Patients with chronic pain conditions
* Patients who have difficulty cooperating or have language barriers
* Patients who do not provide written consent
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From the date of ethics committee approval, patients diagnosed with acute appendicitis in the emergency department and determined to undergo definitive surgery following general surgical consultation: patients with suspected acute appendicitis based on history, physical examination, laboratory tests, and Alvarado score calculation, and confirmed by ultrasound (USG) and/or contrast/non-contrast abdominal CT scans.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 1 year after study start date
  Determination of whether TAP-ESP block reduces the need for opioids in the management of acute appendicitis pain in the emergency department.

SECONDARY OUTCOMES:
Secondary Outcome | 1 year after study start date
  Evaluation of the effectiveness of multimodal pain control for acute appendicitis pain in the emergency department across different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Burak Erdem, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)